CLINICAL TRIAL: NCT06565169
Title: Improving Primary Care Clinician's Advance Care Planning Alzheimer's Disease and Related Dementias
Brief Title: Improving PCP Advance Care Planning for People With ADRD
Acronym: AD-ACP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Chrissy Kistler, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY23080154; 24-0203 (Other: University of North Carolina, Chapel Hill); 1R01AG083828 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-21 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Dementia; Alzheimer's Disease (Incl Subtypes); Aging
Keywords: Advance Care Planning; Primary Care; Goals of Care; Communication
MeSH Terms: conditions — Alzheimer Disease; Dementia; Communication | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and all personnel involved in the outcomes assessment will remain masked to study arm assignment until the end of the study, while the UNC site co-investigators will deliver training and feedback reports to intervention sites and will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Advance Care Planning Training (Experimental): 1. Dementia-specific education: Stage-specific findings and challenges, including AD/ADRD staging, capacity assessment, symptom burden, hospice guidelines, etc - 10-minute didactics, delivered via video conferencing and via the website
  2. ACP communication skills: Context-specific skills and tips on how to slow down, set the communication stage, active listening, respect for personhood and cultural norms, and common, useful language to prepare patients and families- 10-minute didactics, delivered via video conferencing and via the website
  3. Clinical implementation support: Coding and billing information for ACP and ACP templates, an action plan for each team member participant, monthly ACP audit-and-feedback to participants, monthly coaching sessions, site champion, refresher sessions, and educational in-services as needed - Resources at the end of the training session, available on the website, monthly feedback reports on ACP practices, periodic coaching
  Interventions: Behavioral: Primary Care Team Advance Care Planning With People with Alzheimer's Disease or a Related Dementia Training
- Care as Usual: No Training (Active Comparator): These primary care teams will not receive the Advance Care Planning training. Clinics randomized to the control arm will have access to voluntary, routine ACP training sessions provided by UNC HEALTH. We will provide the control clinics summary reports of their ACP practice outcomes at the end of the 18-month follow-up period, which can be used in future practice improvement efforts.
  Interventions: Behavioral: Care as Usual

INTERVENTIONS:
Behavioral: Primary Care Team Advance Care Planning With People with Alzheimer's Disease or a Related Dementia Training — Included in arm/group descriptions
  Other Names: AD-ACP
  Arms: Intervention: Advance Care Planning Training
Behavioral: Care as Usual — Included in arm/group descriptions
  Arms: Care as Usual: No Training

SUMMARY:
This study will test the Dementia Advance Care Planning (AD ACP) Toolkit intervention to usual care in facilitating goals of care (GOC) discussions between People Living with Dementia (PLwD) and primary care team members over an 18-month period. The primary outcome is to assess the frequency and quality of GOC discussions with PLwD. Secondary outcomes include the identification of preferred surrogates, assessment of decisional capacity, and the completion of portable ACP orders. This randomized clinical trial aims to determine if the AD ACP Toolkit can enhance ACP practices and improve care planning outcomes for PLwD compared to the standard care approach.

DETAILED DESCRIPTION:
This project will test an advance care planning (ACP) toolkit for primary care teams caring for patients living with Alzheimer's Disease and related dementias (AD/ADRD) in a cluster randomized control trial. In 20 primary clinics, the advance care planning practices, including goals of care discussions will be examined as the primary outcome, with secondary outcomes including health care utilization, and implementation outcomes. The AD ACP intervention will be tested to determine whether it can enable primary care teams to better conduct goals of care (GOC) discussions more efficiently and thus increase the number of GOC discussions held as compared to controls. The AD ACP Toolkit will be delivered to 10 intervention primary care clinics and usual care to 10 control clinics using a computerized case-finding algorithm within a large integrated health care system. The primary aim is to conduct a trial comparing the AD ACP Toolkit to usual care on GOC discussions and other ACP measures. The second aim is to examine the 18-month healthcare utilization outcomes for all PLwD with >50% 5-year mortality risk between intervention and control. Secondary analyses will be conducted to examine outcomes by key patient and team characteristics. Lastly (aim 3), implementation will be assessed via surveys in the intervention clinics followed by interviews to explain variations in those outcomes. This work will improve how to incorporate ACP approaches for aging-related conditions by primary care teams and may be adaptable to other outpatient specialties such as oncology or cardiology.

ELIGIBILITY:
Inclusion Criteria:

Primary care team member (PCTM) eligibility:

* Must be an MD/APP, employed at a primary care clinic within UNC HEALTH clinics with ≥60 PLwD encounters per year, who sees older adult patients, along with their associated nurses and social workers.
* Eligibility for training with AD ACP Toolkit will include the above and the provision of care at an intervention clinic.
* For Aim 3, only the trained intervention site primary care team members will be eligible for the implementation surveys or the interviews.

PLwD eligibility:

* Must be a PLwD age 65 years or older seen by either the intervention or control sites' primary care teams' MD/APP in the 18-month intervention window for Aim 1.
* PLwD will be eligible only after we confirm the presence of the AD/ADRD diagnosis.
* All PLwD with a ≥50% 5-year all-cause mortality risk seen by the PCTM MD/APP over the 18-month intervention period will be eligible for the healthcare utilization analyses in Aim 2.

Exclusion Criteria:

Primary care team member exclusion criteria:

* We will exclude primary care team members who do not care for older adults (e.g. pediatricians or lactation nurses), are employed at geriatric specialty or dementia specialty clinics, or are without a primary care panel (e.g., only urgent care).

PLwD exclusion criteria:

* Patients will be excluded if they have not been seen in the past 18 months by their primary care team, or if they do not have a diagnosis of ADRD.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Goals of Care Discussions | 18 months
  Presence of a documented Goals of Care (GOC) discussion between the primary care team member and the Person Living with Dementia (PLwD) or their surrogate decision-maker. Medical record documentation of discussion must include a) communication about dementia stage or prognosis AND b) decision-making for at least one major treatment: CPR/mechanical ventilation, hospitalization, treatments for infections, artificial/feeding/hydration, OR hospice.

SECONDARY OUTCOMES:
Surrogate Decision-Maker | 18 months
  Choice of a surrogate decision-maker for the PLwD documented in the medical record.
Decision-Making Capacity | 18 months
  Assessment and report of decision-making capacity for the PLwD documented in the medical record.
Portable Advance Care Planning (ACP) Orders | 18 months
  Completion of portable ACP orders using a state-approved DNR or POLST form documented in the medical record.
Prognosis Discussion | 18 months
  Discussion of prognosis or future medical complications of Alzheimer's Disease/Alzheimer's Disease and Related Dementias (AD/ADRD) between the primary care team member and the PLwD or their surrogate decision-maker documented in the medical record.
Hospital Transfers | 30 months
  Number of emergency room visits and hospital admissions.
Adoption | 30 months
  The percentage of active users at each clinic who have completed at least one training of either type
Length-of-Stay | 30 months
  Duration of hospitalizations from day of admission to day of discharge.
Palliative Care Referral | 30 months
  Percent of PLwD with a referral order to Palliative Care in the medical record.
Hospice Referral | 30 months
  Percent of PLwD with a referral order to Hospice in the medical record.
Goal-concordant care | 30 months
  Number of documented code status and health care proxy in the medical records
Acceptability | 6 months after provider training
  Scores of Organizational Readiness to Implementing Change (ORIC) - range 12-60 with higher scores indicating greater organizational readiness
Appropriateness | 30 months
  Scores of Intervention Appropriateness Measure (IAM) - range 4-20 with higher scores indicating greater appropriateness
Feasibility | 30 months
  Scores of Feasibility of Intervention Measure (FIM) - range 4-20 with higher scores indicating greater feasibility
Fidelity | 30 months
  Scores of primary care team members on post-intervention quizzes, participation in clinic-level and primary care team member-level ACP audit-and-feedback, refresher sessions and in-services, periodic coaching from the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Christine E. Kistler, MD, MASc, Principal Investigator — University of Pittsburgh, Department of Medicine, Division of Geriatric Medicine; Laura C. Hanson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. In addition, every attempt will be made to publish results in peer-reviewed journals. Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 9 months after publication and indefinitely
Access Criteria: Data may be requested to achieve aims in an approved proposal by contacting the PI and The North Carolina Translational and Clinical Science Institue (TraCS)
URL: https://tracs.unc.edu/

REFERENCES:
- [Background] Levine DM, Linder JA, Landon BE. Characteristics and Disparities among Primary Care Practices in the United States. J Gen Intern Med. 2018 Apr;33(4):481-486. doi: 10.1007/s11606-017-4239-z. Epub 2017 Dec 4. PMID 29204975
- [Background] Ernecoff NC, Wessell KL, Gabriel S, Carey TS, Hanson LC. A Novel Screening Method to Identify Late-Stage Dementia Patients for Palliative Care Research and Practice. J Pain Symptom Manage. 2018 Apr;55(4):1152-1158.e1. doi: 10.1016/j.jpainsymman.2017.12.480. Epub 2017 Dec 27. PMID 29288881
- [Background] Kistler CE, Beeber AS, Winzelberg GS, Gabriel SL, Wretman CJ, Hanson LC. Evaluation of a Training Toolkit to Improve Clinicians' Skills for Dementia Advance Care Planning. J Palliat Med. 2021 Aug;24(8):1183-1190. doi: 10.1089/jpm.2020.0638. Epub 2021 Jan 5. PMID 33400605
- [Background] Drabo EF, Barthold D, Joyce G, Ferido P, Chang Chui H, Zissimopoulos J. Longitudinal analysis of dementia diagnosis and specialty care among racially diverse Medicare beneficiaries. Alzheimers Dement. 2019 Nov;15(11):1402-1411. doi: 10.1016/j.jalz.2019.07.005. Epub 2019 Sep 4. PMID 31494079
- [Background] Lund JL, Kuo TM, Brookhart MA, Meyer AM, Dalton AF, Kistler CE, Wheeler SB, Lewis CL. Development and validation of a 5-year mortality prediction model using regularized regression and Medicare data. Pharmacoepidemiol Drug Saf. 2019 May;28(5):584-592. doi: 10.1002/pds.4769. Epub 2019 Mar 19. PMID 30891850
- [Background] Kelley AS, McGarry K, Fahle S, Marshall SM, Du Q, Skinner JS. Out-of-pocket spending in the last five years of life. J Gen Intern Med. 2013 Feb;28(2):304-9. doi: 10.1007/s11606-012-2199-x. Epub 2012 Sep 5. PMID 22948931
- [Background] Dinnen T, Williams H, Yardley S, Noble S, Edwards A, Hibbert P, Kenkre J, Carson-Stevens A. Patient safety incidents in advance care planning for serious illness: a mixed-methods analysis. BMJ Support Palliat Care. 2019 Aug 28;12(e3):e403-10. doi: 10.1136/bmjspcare-2019-001824. Online ahead of print. PMID 31462421
- [Background] Boustani M, Peterson B, Hanson L, Harris R, Lohr KN; U.S. Preventive Services Task Force. Screening for dementia in primary care: a summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Jun 3;138(11):927-37. doi: 10.7326/0003-4819-138-11-200306030-00015. PMID 12779304
- [Background] Xie J, Brayne C, Matthews FE; Medical Research Council Cognitive Function and Ageing Study collaborators. Survival times in people with dementia: analysis from population based cohort study with 14 year follow-up. BMJ. 2008 Feb 2;336(7638):258-62. doi: 10.1136/bmj.39433.616678.25. Epub 2008 Jan 10. PMID 18187696
- [Background] Tinetti ME, McAvay GJ, Murphy TE, Gross CP, Lin H, Allore HG. Contribution of individual diseases to death in older adults with multiple diseases. J Am Geriatr Soc. 2012 Aug;60(8):1448-56. doi: 10.1111/j.1532-5415.2012.04077.x. Epub 2012 Jun 26. PMID 22734792
- [Background] Bernstein A, Rogers KM, Possin KL, Steele NZR, Ritchie CS, Kramer JH, Geschwind M, Higgins JJ, Wohlgemuth J, Pesano R, Miller BL, Rankin KP. Dementia assessment and management in primary care settings: a survey of current provider practices in the United States. BMC Health Serv Res. 2019 Nov 29;19(1):919. doi: 10.1186/s12913-019-4603-2. PMID 31783848